CLINICAL TRIAL: NCT01693185
Title: Remifentanil Only vs. Combination Group Midazolam + Meperidine During Elective Colonoscopy
Brief Title: Remifentanil Only vs. Midazolam and Meperidine During Elective Colonoscopy
Acronym: remifentanil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH1160048
Record Dates: First submitted 2012-09-17; First posted 2012-09-26 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Diagnostic Colonoscopy Screening
Keywords: colonoscopy; remifentanil; midazolam; meperidine
MeSH Terms: interventions — Remifentanil; Midazolam; Meperidine; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Experimental): remifentanil of 0.04 mcg/kg/min with placebo (for midazolam) and placebo (for meperidine)
  Interventions: Drug: Remifentanil; Drug: placebo (for midazolam); Drug: placebo (for meperidine)
- midazolam and meperidine (Active Comparator): a bolus midazolam of 0.03 mg/kg a bolus meperidine of 1.0 mg/kg placebo (for remifentanil)
  Interventions: Drug: Midazolam; Drug: Meperidine; Drug: placebo (for remifentanil)

INTERVENTIONS:
Drug: Remifentanil — continuous infusion 0.4 mcg/kg/min
  Other Names: Ultiva
  Arms: Remifentanil
Drug: Midazolam — bolus injection
  Other Names: dormicum
  Arms: midazolam and meperidine
Drug: Meperidine — bolus injection for 30 sec 1.0 mg/kg
  Other Names: Pethidine Injection
  Arms: midazolam and meperidine
Drug: placebo (for remifentanil) — normal saline mimic diluted remifentanil
  Other Names: normal saline
  Arms: midazolam and meperidine
Drug: placebo (for midazolam) — normal saline mimic to midazolam injection
  Other Names: normal saline
  Arms: Remifentanil
Drug: placebo (for meperidine) — normal saline mimic meperidine injection
  Other Names: normal saline
  Arms: Remifentanil

SUMMARY:
The aim of the present study is to compare patient's recovery times after elective colonoscopy employing remifentanil only vs conventional combination of midazolam and meperidine

DETAILED DESCRIPTION:
A regimen with combined administration of midazolam and meperidine has been widely used and provides quite satisfactory sedation as well as analgesia during colonoscopy. However, the relatively long duration of midazolam and meperidine often prolongs the recovery time after colonoscopy and delays discharge time. (Reimann FM , Samson U , Derad I et al. Synergistic sedation with low-dose midazolam and propofol for colonoscopies . Endoscopy 2000 ; 32 : 239 - 44).

Remifentanil, an ultra-short-acting opioid, provides excellent pain control during colonoscopy and its rapid onset and offset times are advantages over other conventional opioids including meperidine, in avoiding prolonged discharge time after the colonoscopy.

A total 54 patients, aged 18-65 years in American Society of Anesthesiologists physical status (ASA PS)1 and 2, scheduled for elective colonoscopy under Monitored Anesthesia Care in a University Hospital, will be recruited after obtaining written informed consent during the patients' first visit to outpatient/inpatient clinic for interview.

Predetermined patient identification numbers (PIN) and enrolment order were placed in sealed envelopes, and all patients were randomly assigned, at recruitment, to the midazolam-meperidine combination (group-MM) or remifentanil alone (group-R). If a patient was excluded during the study, the following patient assumed the status of the excluded patient.

Patients are allocated into one of two groups, Group 1 and Group 2 (27 patients each) according to the PIN at the recruitment.

The exclusion criteria were as follows: refusal or inability to provide written informed consent, age <19 years, pregnancy, previous history of large bowel surgery, a psychiatric disorder, an addictions to opiates or sedatives, a previous history of adverse events to any drug used in the present study, and performance of any additional diagnostic procedure after completion of colonoscopy.

All colonoscopic procedure is going to be performed by one Gastroenterologist (endoscopist).

On arriving in the endoscopy room, supplemental oxygen (2 L/min) was given through the mouth and both nostrils via a specially designed nasal prong which could monitor the end-tidal CO2 (ETCO2) level.

Before drug administration, the basal values of mean blood pressure (MBP), heart rate (HR), peripheral O2 saturation (SpO2), respiratory rate (RR), end-expiratory CO2 level (ETCO2), and the bispectral index (BIS), were recorded by a single observer, who also monitored these values every 5 min during entire colonoscopy procedures.

Supplemental oxygen (3 L/min) is given through nasal prong with capnography transducer in all patients.

Two min before the colonoscopy procedure, a bolus midazolam of 0.03 mg/kg with a bolus meperidine of 1.0 mg/kg are given intravenously over 60 sec in Group 1 or those of comparable amount of diluted remifentanil 0.4 mcg/kg are given in Group 2 at the colonoscopy room, and a continuous infusion of diluted remifentanil of 0.04 mcg/kg/min is followed in Group 2 or that of comparable amount of normal saline (placebo) is followed in Group 1.

The patients are asked to rate the degree of pain and distress (reverse satisfaction) by a 100 mm Visual analogue scale (VAS; 0 = minimum, 100 = maximum) just after passing the scope, during the scope, just after the completion of the colonoscopy and at the discharge from the recovery unit.

After colonoscopy, the patients are transferred to the recovery unit and evaluated every 5 min until ready for discharge from the 30 min stay in the recovery unit.

The patients are considered recovered if when they achieved an Aldrete score of 10 (Aldrete JA , Kroulik D . A postanesthetic recovery score. Anesth Analg 1970; 49: 924 - 34), have stable vital signs, are able to tolerate oral fluids, have no nausea, vomiting, or itching, and can walk unaided.

Assessment of readiness to ambulate is made by a blinded observer who remained with the patient for the duration of recovery unit stay.

The observer is instructed that the patients are required to walk as if they were leaving the recovery unit unescorted.

Aldrete score, patient pain and satisfaction (distress score) were determined every 5 min during colonoscopy and after colonoscopy up to 30 min. Time for achieving Aldrete score 10, patient's degree of pain, patient's satisfaction during and after colonoscopy, patient's ability to recall the explanations and instructions given during and before colonoscopy are determined and compared.

Aldrete score Respiration: Able to take deep breath and cough = 2, Dyspnea/shallow breathing = 1, Apnea = 0 O2 saturation: Maintains > 92% on room air =2, Needs O2 inhalation to maintain O2 saturation > 90% =1 , O2 saturation < 90% even with supplemental oxygen =0 Consciousness: Fully awake= 2, Arousable on calling = 1, Not responding = 0 Circulation: BP +/- 20 mm Hg preop =2, BP +/- 20-50 mm Hg preop =1, BP +/- 50 mm Hg preop =0 Activity: Able to move 4 extremities = 2, Able to move 2 extremities = 1, Able to move 0 extremities = 0

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-65 years
* American Society of Anesthesiologists physical status (ASA PS) 1-2
* Patients scheduled for elective colonoscopy under Monitored Anesthesia Care in a University Hospital
* Patients who signed on written informed consent.

Exclusion Criteria:

* The exclusion criteria are refusal or inability to provide written informed consent
* Age < 18 years
* Pregnancy
* Previous large bowel surgery
* Psychiatric disorders
* History of addiction to opiates and / or sedatives, and previous adverse reaction to any drug used in the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Predetermined patient identification numbers and enrolment order were placed in sealed envelopes, and all patients were randomly assigned, at recruitment, to the midazolam-meperidine combination (group-MM) or remifentanil alone (group-R). If a patient was excluded during the study, the following patient assumed the status of the excluded patient.
Pre-assignment Details: The exclusion criteria were applied. If a patient was excluded after recruitment and enrollment into the study, the following new patient assumed the status of the excluded patient.
Period: Overall Study
Arm/Group | Remifentanil | Midazolam and Meperidine
Started | 27 | 33
Completed | 27 | 27
Not Completed | 0 | 6
Not completed — diagnostic procedure after colonoscopy | 0 | 6

BASELINE CHARACTERISTICS:
Population: Patients with ASA PS class 1 or 2 undergoing elective colonoscopy under monitored anesthesia care
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Midazolam and Meperidine | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.7) | 53.0 (10.7) | 54.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Recovery Time
Description: Time from completing the colonoscopy to achieving Aldrete score 10 in the recovery unit
  Aldrete score
  * Respiration: Able to take deep breath and cough = 2, Dyspnea/shallow breathing = 1, Apnea = 0
  * O2 saturation: Maintains > 92% on room air =2, Needs O2 inhalation to maintain O2 saturation > 90% =1 , O2 saturation < 90% even with supplemental oxygen =0
  * Consciousness: Fully awake= 2, Arousable on calling = 1, Not responding = 0
  * Circulation: BP +/- 20 mm Hg preop =2, BP +/- 20-50 mm Hg preop =1, BP +/- 50 mm Hg preop =0
  * Activity: Able to move 4 extremities = 2, Able to move 2 extremities = 1, Able to move 0 extremities = 0
  To estimate the required sample size, we conducted a pilot study to measure the recovery of 10 patients in each of groups-MM and -R before the present study. The means and standard deviations were 22.5 ± 9.5 and 7.5 ± 9.2 min respectively. We wished to be able to distinguish a difference of 7.5 min, thus half of the observed difference.
Time Frame: every 5 minutes after completing colonoscopy up to 30 min
Measure: Median (Inter-Quartile Range); unit: minute
Arm/Group | Remifentanil | Midazolam and Meperidine
Number analyzed (Participants) | 27 | 27
minute | 0 [0 to 10] | 30 [15 to 30]
Statistical Analysis 1: Comparison: Remifentanil vs Midazolam and Meperidine; Recovery time in patients administered remifentanil alone will be significantly shorter than that in patients administered midazolam-meperidine combination for colonoscopy; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — We wished to be able to distinguish a difference of 7.5 min,

2. Secondary Outcome: Participants Assumed to Feel Frequent Pain
Description: patients sound "Ah" at feeling pain during colonosocpy: if a patients sounds "Ah" > 6 times, the patient was assumed to feel frequent pain.
Time Frame: during and after colonoscopy
Measure: Number; unit: participants
Arm/Group | Remifentanil | Midazolam and Meperidine
Number analyzed (Participants) | 27 | 27
participants | 4 | 7

3. Secondary Outcome: Bispectra Lindex Score
Description: Bispectral index (BIS) score 0-100 maximal sedation=0, maximal sedation=100
Time Frame: every 5 min during and after colonoscopy
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Remifentanil | Midazolam and Meperidine
Number analyzed (Participants) | 27 | 27
units on a scale | 92 [85 to 96] | 84 [80 to 87]

4. Secondary Outcome: Patient's Distress Score
Description: patients' distress in visual analogue scale 100 mm minimal distress=0, maximal distress=100
Time Frame: 5 min after the end of colonoscopy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remifentanil | Midazolam and Meperidine
Number analyzed (Participants) | 27 | 27
units on a scale | 37 [30 to 43] | 30 [30 to 30]

5. Secondary Outcome: Endoscopist Satisfaction
Description: endoscopist's satisfaction after colonoscopy in visual analogue scale 100 mm
Time Frame: 5 min after the colonoscopy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remifentanil | Midazolam and Meperidine
Number analyzed (Participants) | 27 | 27
units on a scale | 5 [5 to 10] | 20 [10 to 20]

6. Secondary Outcome: Indigence of Patient's Recall
Description: The numbers of patients who recalled instructions and explanations given during colonoscopy
Time Frame: after colonoscopy
Measure: Number; unit: participants
Arm/Group | Remifentanil | Midazolam and Meperidine
Number analyzed (Participants) | 27 | 27
participants | 27 | 13

ADVERSE EVENTS:
Time Frame: during and after colonosocpy, up to 30 min
Description: incidence (number of patients) of pulse oximetry < 90% during colonoscopy during and after colonoscopy
Arm/Group | Remifentanil | Midazolam and Meperidine
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No